CLINICAL TRIAL: NCT07060183
Title: Aortic Valve Replacement for Moderate Aortic Stenosis With Left Ventricular Decompensation Early Feasibility Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Dermed Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Moderate Aortic Stenosis AVR
Record Dates: First submitted 2023-04-25; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Moderate Aortic Valve Stenosis
Keywords: aortic; stenosis; valve; decompensation; moderate
MeSH Terms: conditions — Constriction, Pathologic; Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Aortic Valve Replacement
  Interventions: Procedure: Ross procedure
- Control (No Intervention): No intervention

INTERVENTIONS:
Procedure: Ross procedure — aortic valve replacement
  Arms: Intervention

SUMMARY:
Obtain safety and effectiveness data to support expansion for aortic valve replacement to include patients with moderate aortic stenosis and left ventricular decompensation.

DETAILED DESCRIPTION:
Single-center prospective study. Subjects with moderate aortic stenosis and left ventricular decompensation will receive aortic valve replacement by the Ross procedure.

ELIGIBILITY:
Inclusion Criteria:

* Moderate aortic stenosis, defined by transthoracic echocardiograph
* Max aortic velocity less than 4.0 m/sec.
* Mean aortic gradient less than 40.0 mmHg.
* 1.0 cm2 < Aortic Valve Area < 1.5 cm2.
* Left ventricular decompensation

Exclusion Criteria:

* Not suitable for the Ross procedure.
* Documented history of cardiac amyloidosis.

Ages: 55 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2027-01 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Composite rates of all-cause mortality or morbidity | 12 months
  Composite rate of all-cause mortality, all-stroke, life threatening or fatal bleeding, acute kidney injury, hospitalization due to procedure-related complication, or valve dysfunction requiring reintervention.

SECONDARY OUTCOMES:
Left ventricular compensation | 12 months
  Improvement in left ventricular function from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Arthur P DeMarzo, Study Director — Dermed Diagnostics, Inc.

IPD SHARING:
Plan to Share IPD: No